CLINICAL TRIAL: NCT03799796
Title: Combining Flash Glucose Monitoring and Online Peer Support to Improve Outcomes in Hispanic Spanish-Speaking People With Type 2 Diabetes
Brief Title: Combining Flash Glucose Monitoring and Online Peer Support to Improve Outcomes in Hispanics With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: La Trobe University (Other)
Responsible Party: Principal Investigator, Michelle Litchman, Assistant Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ADC-SRR-IIS-18-23
Record Dates: First submitted 2019-01-09; First posted 2019-01-10 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: flash glucose monitoring; online peer support; Hispanic; Spanish-Speaking
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Flash Glucose Monitoring with Online Peer Support (Experimental): Pre-Test-Post-Test
  Interventions: Behavioral: Flash Glucose Monitoring with Online Peer Support

INTERVENTIONS:
Behavioral: Flash Glucose Monitoring with Online Peer Support — Hispanic Adults who are Spanish-Speaking with type 2 diabetes who are not using insulin will be asked to use flash glucose monitoring and to sign up for an moderated online peer support group where they can ask questions and share progress.
  Other Names: Abbott Freestyle Libre

SUMMARY:
Currently, Hispanic Spanish-speaking individuals are not receiving culturally appropriate diabetes care. Lack of knowledge impacts several areas of type 2 diabetes (T2D) management, including healthy eating and being physically active in Hispanic Spanish-speaking individuals. Use of diabetes technology is on the rise, however, many technologies do not provide Spanish-language options. A flash glucose monitoring (FGM) system is now available in both English and Spanish. Research suggests that use of FGM results in improved clinical outcomes. Furthermore, increased number of FGM scans are associated with improved clinical outcomes such as decreased A1C and improvements in BG time in range. Our preliminary work indicates that Hispanics (1) are willing to use diabetes technology, such as FGM, if it supports Spanish language and (2) in English-speaking populations, but not specific to the Hispanic Spanish-speaking population, FGM supports biobehavioral change. Further, our work, and the work of others, indicate Hispanic individuals desire for peer interactions to relate and understand the variables that impact T2D. Interaction with online peer support communities is associated with increased knowledge, receipt of emotional support, and improved glycemic levels. These results suggest that education and support to increase use and understanding of FGM will lead to improved clinical and behavioral outcomes.

DETAILED DESCRIPTION:
Currently, Hispanic Spanish-speaking individuals are not receiving culturally appropriate diabetes care. Lack of knowledge impacts several areas of type 2 diabetes (T2D) management, including healthy eating and being physically active in Hispanic Spanish-speaking individuals. Use of diabetes technology is on the rise, however, many technologies do not provide Spanish-language options. A flash glucose monitoring (FGM) system is now available in both English and Spanish. FGM involves wearing an interstitial glucose sensor that is placed on the upper arm and a reader. When an individual wants to check their glucose level, they waive or scan the reader over their sensor and a glucose history, current glucose level, and projected glucose trend is displayed. Research suggests that use of FGM results in improved clinical outcomes. Furthermore, increased number of FGM scans are associated with improved clinical outcomes such as decreased A1C and improvements in BG time in range. Our preliminary work indicates that Hispanics (1) are willing to use diabetes technology, such as FGM, if it supports Spanish language and (2) in English-speaking populations, but not specific to the Hispanic Spanish-speaking population, FGM supports biobehavioral change. Further, our work, and the work of others, indicate Hispanic individuals desire for peer interactions to relate and understand the variables that impact T2D. Interaction with online peer support communities is associated with increased knowledge, receipt of emotional support, and improved glycemic levels. These results suggest that education and support to increase use and understanding of FGM will lead to improved clinical and behavioral outcomes.

Little is known about the uses, benefits, and limitations of online peer support in the context of learning how to use diabetes technology, such as FGM. Hispanic, Spanish speaking individuals are at high risk for T2D and associated morbidity and mortality. Hispanics are more likely to die from diabetes compared to Caucasian counterparts. The investigators propose to address gaps in diabetes care for Hispanic individuals by conducting a pilot trial of an online peer support intervention using an online peer facilitator to augment the use of FGM. The online peer facilitator will be Hispanic and bilingual in English and Spanish with substantial knowledge of diabetes and FGM. Our intervention is culturally appropriate to address the biobehavioral and biopsychosocial needs of Hispanic individuals. The investigators anticipate the additional support provided by the online peer facilitator will encourage healthy eating habits and physical activity behaviors in Hispanic individuals with T2D. Our research team is experienced with community-based participatory research in both diabetes online peer support communities and Hispanic populations using technology to support T2D.

Examining online peer support communities to augment diabetes care in Hispanic Spanish speaking individuals is a promising, exciting, and innovative area of research that has not yet been explored. This proposed study contains several novel components. First, using online peer support communities is low-cost and easily accessible, making this intervention more translatable in the clinical setting while adding to the toolkit that already exists for diabetes care. Second, using FGM in a population not using insulin is forward thinking. Empowering people with their own glucose data, early in the course of their diabetes, may change the trajectory of diabetes management. The research team received PCORI pipeline-to-proposal funding (tiers I-III) to develop a research question via a community advisory board (CAB) in partnership with the diabetes online peer support community. The CAB included researchers, clinicians, and people with diabetes, both English and Spanish speaking. This study will address important questions identified by people affected by diabetes.

Aim 1 Explore the relationship between engagement in an online peer support intervention with clinical and behavioral outcomes in Hispanic, Spanish speaking individuals with T2D using flash glucose monitoring for 12 weeks

Method. A one group, pre-post evaluation of Hispanic, Spanish speaking individuals (N=43) recruited from a health center in Utah.

Primary outcome: Time-in-range (average glucose level and number of minutes in 70mg/dl-180mg/dl in last 10 days of the study minus average glucose level and number of minutes in 70mg/dl-180mg/dl for 10 days baseline) between baseline and 12 weeks.

Secondary outcomes: Change in A1C from baseline to 12 weeks. Online peer support engagement (measured by survey and Facebook activity), Frequency of FGM scans. Change in self-reported self-management behaviors, self-efficacy and quality of life between baseline and 12 weeks.

Hypothesis. Increased engagement in the online peer support intervention will be associated with improved clinical, behavioral and psychosocial outcomes after 12 weeks of FGM.

Aim 2. Evaluate the acceptability and feasibility of an online peer support intervention for Hispanic Spanish speaking individuals with T2D to learn how to use flash glucose monitoring to make changes to meal and activity choices.

Method. Qualitative and quantitative analysis for measures of use of and satisfaction with flash glucose sensors, eligible participant acceptance of flash glucose sensors, and dropout rates, including causes for drop out, and online peer support engagement through platform analytics. A semi-structured interview will be conducted with participants at the end of the intervention explore their experiences during engagement with the online peer support community.

Hypothesis. Online peer support engagement will be associated with satisfaction with FGM and number of daily scans.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥21 years
* Self-report as Hispanic
* Able to communicate in Spanish
* Clinical diagnosis of T2D and HbA1c ≥8% per clinic records
* Willing to wear a flash glucose monitor for 12 weeks
* Access to the internet and willing to engage in an online peer support community
* Willing to avoid Vitamin C 500 mg and Aspirin 325 mg or greater daily
* Not using insulin

Exclusion Criteria:

* Non-Spanish speaking
* Using insulin
* Already using a continuous glucose monitor or flash glucose monitor in previous 6 months
* Participation in other diabetes clinical trials
* Alcohol or drug abuse/dependency
* Severe illness (physical or mental health), cognitive impairment, high dose steroids, hospitalized more than 2 times in past 12 months or other impairment that would, in the opinion of the investigators, interfere with ability to complete the study
* Uncorrected hearing or vision impairment
* Life expectancy <6 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-01-06 (Actual); Primary Completion 2020-07-27 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Time-in-Range | 12 weeks
  Average glucose level and number of minutes spent between 70-180 mg/dL

SECONDARY OUTCOMES:
A1C | 12 weeks
  Glycosylated hemoglobin
Online peer support engagement | 12 weeks
  Survey, Activity in online peer support group

CONTACTS AND LOCATIONS:
Overall Officials: Michelle L Litchman, PhD, FNP-BC, Principal Investigator — University of Utah College of Nursing
Locations (1):
- University of Utah College of Nursing, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data can be shared upon request.

REFERENCES:
- [Derived] Ng AH, Greenwood DA, Iacob E, Allen NA, Ferrer M, Rodriguez B, Litchman ML. Examining a Continuous Glucose Monitoring Plus Online Peer Support Community Intervention to Support Hispanic Adults With Type 2 Diabetes: Protocol for a Mixed Methods Feasibility Study. JMIR Res Protoc. 2022 Feb 24;11(2):e31595. doi: 10.2196/31595. PMID 35200153